CLINICAL TRIAL: NCT04446611
Title: Clinical Study of STI Screening to Prevent Adverse Birth and New-born Outcomes
Brief Title: Clinical Study of STI Screening to Prevent Adverse Birth and New-born Outcomes (Philani Ndiphile)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Professional Development (Pty) Ltd (Other)
Collaborators: University of Southern California (Other); National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Cape Town (Other); University of Alabama at Birmingham (Other); Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: R01AI149339 (NIH); R01AI149339 (NIH)
Record Dates: First submitted 2020-04-15; First posted 2020-06-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Sexually Transmitted Infection; HIV/AIDS; Cost-effectiveness; Birth Outcomes; Vaginal Microbiome; Neisseria Gonorrhoeae; Chlamydia Trachomatis; Trichomonas Vaginalis; Antenatal Care; Pregnancy
Keywords: Sexually transmitted infection; Neisseria gonorrhoeae; Chlamydia trachomatis; Trichomonas vaginalis; Antenatal care; HIV/AIDS; Birth outcomes; South Africa; Vaginal microbiome; Pregnancy; Diagnostic testing
MeSH Terms: conditions — Sexually Transmitted Diseases; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The intervention will incorporate diagnostic testing using the Xpert® platform with same-day treatment for Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis infection at first ANC (aim 1 and 2) with either a test-of-cure (arm 1) or 30 weeks repeat testing as follow-up (arm 2) compared to the standard of care (arm 3), i.e. syndromic management as per the South African guidelines. It is thus a 3-arm (1:1:1) control trial with additional components of vaginal microbiome analysis, economic evaluation and qualitative insights.
Masking Description: The allocation of study arm is concealed to study staff during randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test at 1st ANC + Test-of-Cure (Treatment 1) (Experimental): Single point-in-time diagnostic screening plus test-of-cure three weeks post-treatment
  Interventions: Diagnostic Test: First antenatal care + test-of-cure
- Test at 1st ANC + 30-34 gestation (Treatment 2) (Experimental): Repeated diagnostic screening at first antenatal care and 30-34 weeks gestation
  Interventions: Diagnostic Test: First antenatal care + week 30-34 gestation (no test-of-cure)
- Syndromic Management (Control) (No Intervention): Syndromic management (standard of care) at every antenatal care visit per South African National Guidelines.

INTERVENTIONS:
Diagnostic Test: First antenatal care + test-of-cure — Single point-in-time molecular point-of-care diagnostic screening and treatment for Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis at first antenatal care visit and infection-specific test-of-cure 3 weeks post-treatment. Women with a positive test-of-cure will be re-treated. As CT/NG is a combined Xpert test, women who present with an incident infection (newly diagnosed infection) will be treated and managed accordingly.
  Arms: Test at 1st ANC + Test-of-Cure (Treatment 1)
Diagnostic Test: First antenatal care + week 30-34 gestation (no test-of-cure) — Repeated molecular point-of-care diagnostic screening and treatment for Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis at first antenatal care visit and at week 30-34 gestation. No test-of-cure will be conducted for women with positive test results; however, additional treatment will be provided to women with persistent/recurrent vaginal discharge.
  Arms: Test at 1st ANC + 30-34 gestation (Treatment 2)

SUMMARY:
This study aims to evaluate different screening strategies to decrease the burden of Neisseria gonorrhoeae (NG), Chlamydia trachomatis (CT) and Trichomonas vaginalis (TV) among pregnant women, and reduce adverse birth outcomes. In turn it aims to evaluate the cost per pregnant woman screened and treated, cost of adverse birth outcomes, and cost-effectiveness per sexually transmitted infection (STI) and disability-adjusted life-year (DALY) averted. Furthermore, this study will incorporate a vaginal microbiome sub-study aimed to investigate the relationship between the vaginal microbiome and persistent Chlamydial infections in pregnant women.

Aim 1 and 2: The intervention includes diagnostic testing at a woman's first antenatal care visit using the Xpert® platform with same-day treatment for Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis infection with either a test-of-cure three weeks post-treatment (arm 1) or a repeat test at 30-34 weeks gestation (arm 2) compared to the standard of care, i.e. syndromic management (arm 3).

Aim 3: Case-control study to investigate role vaginal microbiome in STI treatment outcomes

DETAILED DESCRIPTION:
Prevalence of STIs is high among pregnant women in South Africa and most infections remain untreated. Untreated infections impact on pregnancy and birth outcomes. Good diagnostic and point-of-care (POC) tests are available, such as the GeneXpert platform. The health impact, cost-effectiveness and approaches to optimization of STI diagnostic screening during pregnancy are unknown.

In order to 1) identify optimal, cost-effective screening strategies that decrease the burden of STIs during pregnancy and reduce adverse birth outcomes, 2) informs evidence to WHO's guidelines to introduce aetiologic STI screening globally and 3) elucidate the role of the vaginal microbiome in STI treatment outcomes, the investigators propose three Specific Aims:

1. Evaluate different screening strategies to decrease the burden of Neisseria gonorrhoeae, Chlamydia trachomatis and Trichomonas vaginalis among pregnant women and reduce adverse birth outcomes
2. Evaluate cost per pregnant woman screened and treated, cost of adverse birth outcomes, and cost-effectiveness per STI and disability-adjusted life-year (DALY) averted
3. Investigate the relationship between the vaginal microbiome and persistent Chlamydial infections in pregnant women

STI screening and treatment for Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis will be offered to HIV-infected and non-infected women (age >18 years) whom present for first antenatal care services. An effectiveness-implementation hybrid type 1 three-arm (1:1:1) randomized controlled trial (RCT), will be employed to evaluate different screening strategies to decrease the burden of Chlamydia trachomatis, Neisseria gonorrhoeae and Trichomonas vaginalis among pregnant women, and reduce adverse birth outcomes.

The costs of the different STI screening strategies relative to control will be estimated based on literature review and performance/implementation characteristics and compared, in addition to the costs of managing adverse birth outcomes. Decision analytic modelling will estimate the cost-effectiveness per STI, and DALY averted (Aim 2).

Depending on the randomization arm, participants will be scheduled to be seen various times throughout pregnancy by the study team; antenatal care visits will be conducted in line with national policy. All post-partum mothers and infants will be asked to be seen at the first post-delivery clinic visit.

ELIGIBILITY:
Inclusion Criteria for pregnant women:

1. Age≥18 years
2. Currently pregnant based on positive urine pregnancy test
3. Attending first ANC visit for current pregnancy
4. Gestational age <20 weeks
5. Agreeing to nurse-collected specimens
6. Resident in Buffalo City Municipality (BCM)
7. Intent to deliver in one of the four midwife obstetric units (MOUs) in BCM

Gestational age will be confirmed via ultrasound

Exclusion Criteria:

1. Planning to relocate during pregnancy or deliver in an MOU outside of BCM
2. Unknown HIV status (e.g. refusal, invalid test result)
3. Currently participating in another ANC/HIV study
4. When the ultrasound confirms ≥20 weeks gestation at first ANC

Inclusion criteria for Neonates:

1) born to mothers that provided informed consent to participate in study, 2) provision of updated verbal consent by mother to collect and test specimens for STIs

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2247 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse birth outcomes among study arms | Recorded within 2 weeks of delivery
  Adverse birth outcomes as defined by a composite measure of preterm birth (born alive before 370/7 weeks gestation) or low birth weight (less than 2500g) as recorded in the maternity case records

SECONDARY OUTCOMES:
Change in STI prevalence (a) between baseline visit and delivery within the experimental arms and (b) between the experimental and control arms by delivery. | Between baseline (first antenatal visit <27 weeks' gestation) and delivery outcome (collected within 2 weeks post-delivery)
  To calculate the relative and absolute change in Chlamydia, Gonorrhea, and Trichomoniasis prevalence. Additionally, generalized estimating equations to test for variation in STI prevalence among study arms will be done, adjusting for potential effect modifiers and confounding variables
Correlation between Bacterial vaginosis-associated vaginal community state types and clearance of Chlamydia infection | Assessed through study completion
  To determine the correlation between Bacterial vaginosis-associated vaginal community state types and chlamydial infection clearance as measured by a positive or negative chlamydial test result no less than three weeks after treatment and thence weekly until a negative Chlamydia test result is recorded.
Incidence of Preterm birth among study arms | At delivery
  The frequency of live births before 37 weeks' gestation, as validated by ultrasound dating at first antenatal visit
Incidence of Low birthweight infants among study arms | Within 2 weeks post-delivery
  The frequency of live births with birth weight < 2500g, as recorded in the maternity case records
Incidence of STI in infants exposed to infection in their mothers | STI testing in mother and infants within 2 weeks post-delivery to a maximum of 6 weeks post-delivery
  Frequency of Chlamydia, Gonorrhoeae, and/or Trichomonas infection among infants born to a mother in whom infection is detected post-delivery
Frequency of fetal loss (miscarriage or stillbirth) among study arms | Assessed through study completion
  Composite frequency of miscarriage (<28 weeks' gestation) or stillbirth (> 28 weeks' gestation) and the individual components, as indicated in the maternal case records

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Medina-Marino, PhD, MPH, Principal Investigator — Foundation for Professional Development; Jeffrey Klausner, MD, MPH, Principal Investigator — USC Keck School of Medicine - University of Southern California
Locations (1):
- Buffalo City Metro, East London, Eastern Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, Analytic Code
Access Criteria: Based on contractual agreement

REFERENCES:
- [Derived] Medina-Marino A, Cleary S, Muzny CA, Taylor C, Tamhane A, Ngwepe P, Bezuidenhout C, Facente SN, Mlisana K, Peters RPH, Klausner JD. Sexually transmitted infection screening to prevent adverse birth and newborn outcomes: study protocol for a randomized-controlled hybrid-effectiveness trial. Trials. 2022 May 24;23(1):441. doi: 10.1186/s13063-022-06400-y. PMID 35610666